CLINICAL TRIAL: NCT05209958
Title: The Effect of Preoperative NLR Level on Epidural Analgesia Application in Thoracotomy
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ersagun Tugcugil, Assoc.Prof., Karadeniz Technical University
Other Study IDs: 2020/66
Record Dates: First submitted 2022-01-10; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: C23.550.767.700; C23.550.470
Keywords: Preemptive Epidural Analgesia, Neutrophil/Lymphocyte Ratio, İnflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with NLR level below 2
  Interventions: Diagnostic Test: Neutrophil Lynphosite ratio
- Group B: Patients with NLR level equal to or above 2
  Interventions: Diagnostic Test: Neutrophil Lynphosite ratio

INTERVENTIONS:
Diagnostic Test: Neutrophil Lynphosite ratio — The patients were divided into 2 groups as NLR level above 2 (Group A) (n:32) and NLR level below 2 (Group B) (n:28).

SUMMARY:
The aim of this study is to investigate the relationship of preoperative Neutrophil/Lymphocyte Ratio (NLR) with postoperative pain and the effect of preoperative NLR level on timing of epidural analgesia in thoracotomy.

DETAILED DESCRIPTION:
The study was conducted prospectively in 60 patients aged 18-75 years, ASA I-III, who underwent thoracotomy. The patients were divided into 2 groups as NLR level above 2 (Group A) (n:32) and NLR level below 2 (Group B) (n:28). Each group was divided into subgroups with equal numbers of Prempative analgesia group and control group. Local anesthetic was administered to the preemptive analgesia group (Group P) 20 minutes before the surgical incision through the epidural catheter, and to the control group (Group K) 20 minutes before the patient was awakened from the epidural catheter. NRS levels and additional analgesia needs were recorded at 2, 4, 8, 12 and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient graded as American Society of Anesthesiologist (ASA) physical status, I, II or III
* Patient subjected to thoracotomy operation

Exclusion Criteria:

Patient having morbid obesity,

* Patient having renal failure,
* Patient having hepatic failure,
* Patient having neuropsychiatric disease,
* Patient allergy to the study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 female and male patients aged 18-75 years, in the ASA I-III risk group, who will undergo elective thoracotomy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
preoperative neutrophil lymphoycte ratio | 24 hours before the operation
  To determine the epidural application with preoperative neutrophil lymphoycte ratio
Postoperative opioid requiremen Postoperative opioid requirement | postoperative first 24 hour
  Postoperative opioid requirement for pain relief

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | postoperative first 24 hour
  Numerical Pain Rating Scale in postoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- KaradenızTU, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No